CLINICAL TRIAL: NCT00570817
Title: Nephrotoxicity Induced by High-Dose Methotrexate Infusions to Children With Malignant Diseases
Brief Title: Prevention of Methotrexate Induced Nephrotoxicity and Prolonged Drug Elimination Time With 12 Hours Prehydration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: ML Jørgensen og Gunnar Hansens Foundation (Unknown); Danish Child Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 20070009; The Danish Data; Protection Agency 2007-41-0014
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-01

CONDITIONS: Methotrexate Induced Nephrotoxicity
Keywords: Methotrexate; Nephrotoxicity; Hydration; Acute lymphoblastic leukemia; Non-Hodgkin's lymphoma; Medulloblastoma; Ependymoma; Prolonged elimination time of methotrexate
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Medulloblastoma; Ependymoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): The child will receive prehydration at the methotrexate infusions in the following order:
  At the 1st methotrexate infusion the child will receive 4 hours prehydration. At the 2nd methotrexate infusion the child will receive 12 hours prehydration. At the 3rd methotrexate infusion the child will receive 4 hours prehydration. At the 4th methotrexate infusion the child will receive 12 hours prehydration. At the 5th methotrexate infusion the child will receive 4 hours prehydration. At the 6th methotrexate infusion the child will receive 12 hours prehydration. At the 7th methotrexate infusion the child will receive 4 hours prehydration. At the 8th methotrexate infusion the child will receive 12 hours prehydration.
  Interventions: Other: 12 hours of prehydration
- 2 (Other): The child will receive prehydration at the methotrexate infusions in the following order:
  At the 1st methotrexate infusion the child will receive 12 hours prehydration. At the 2nd methotrexate infusion the child will receive 4 hours prehydration. At the 3rd methotrexate infusion the child will receive 12 hours prehydration. At the 4th methotrexate infusion the child will receive 4 hours prehydration. At the 5th methotrexate infusion the child will receive 12 hours prehydration. At the 6th methotrexate infusion the child will receive 4 hours prehydration. At the 7th methotrexate infusion the child will receive 12 hours prehydration. At the 8th methotrexate infusion the child will receive 4 hours prehydration.
  Interventions: Other: 12 hours of prehydration

INTERVENTIONS:
Other: 12 hours of prehydration — 12 hours of prehydration with an infusion rate of 150 ml/m2/hour with a solution of 5% glucose with 40 mmol sodium bicarbonate/L and 20 mmol potassium chloride/L.

SUMMARY:
Infusions with high-dose methotrexate 5 g/m2 or 8 g/m2 are used to treat children with acute lymphoblastic leukemia (ALL), non-Hodgkin's lymphoma, medulloblastoma and ependymoma. Methotrexate is primarily excreted unchanged by the kidney where it can course acute kidney damage resulting in prolonged time of excretion of the drug. Our main hypothesis is that 12 hours of intravenous hydration before the methotrexate infusion is more efficacious in preventing methotrexate induced kidney damage compared to four hours of hydration.

DETAILED DESCRIPTION:
Infusions with high-dose methotrexate 5 g/m2 or 8 g/m2 are according to the protocol of the Nordic Association for Pediatric Hematology and Oncology 2000 (NOPHO-2000) used to treat children with acute lymphoblastic leukemia (ALL). Treatment with methotrexate 5 g/m2 is also used to treat children with non-Hodgkin lymphoma, medulloblastoma and ependymoma. Methotrexate is primarily excreted unchanged by the kidney where it can course acute nephrotoxicity resulting in prolonged elimination time of the drug. Data from a 10 years retrospective investigation at our pediatric unit show, that in spite of urine alkalinization and intensive hydration the elimination of methotrexate is prolonged in 20-50% of the infusions. The long exposure of a high serum methotrexate concentration is associated with an increased frequency of mucositis and bone marrow suppression. Further more the need of rescue with folic acid is problematic, because it is possibly that it can result in a higher risk of relapse of ALL (Leukemia 2006; Skarby TV). Most ALL protocols prescribe prehydration of 2-6 hours before initiation of the methotrexate infusion and it has never been investigated in a randomized controlled trail if a longer time of prehydration can prevent nephrotoxicity and reduce the risk of prolonged elimination. In our pediatric unit the prehydration is given with a rate of 150 ml/m2/hour with a solution of 5% glucose with 40 mmol sodium bicarbonate/L and 20 mmol potassium chloride/L.

Our main hypothesis is that 12 hours of prehydration is more efficacious in preventing methotrexate induced nephrotoxicity compared to four hours of prehydration. A child enrolled in the study will before half of the methotrexate infusions receive 12 hours of prehydration and before the other half it will receive four hours of prehydration.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 and 21 years at the diagnosis of ALL
* Treatment with high-dose methotrexate 5 g/m2 or 8 g/m2 according to the protocol "Nordic Association for Pediatric Hematology and Oncology 2000 (NOPHO-2000)" or the new protocol (NOPHO-2008) to which enrolment begin approx. January 2009.
* Treatment with high-dose methotrexate 5 g/m2 according to the protocol "Treatment Protocol for T-Cell and B-Precursor Cell Lymphoblastic Lymphoma 2002 of the European Inter-group Co-operation on Childhood Non-Hodgkin-Lymphoma (EICNHL)"
* Treatment of medulloblastoma and ependymoma with high-dose methotrexate 5 g/m2 according to the protocol: "(HIT2000)Hirntumorprotokoll der Hrbeitsgruppe für Hirntumoren" from Deutsche Gesellschaft für Pädiatrische Onkologie und Hämatologie (GPOH).

Exclusion Criteria:

* Patient or parents not willing to give consent.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2007-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Prolonged methotrexate elimination time, defined by serum methotrexate concentrations: > 3,0 micromol/L at 36 hours; > 1,0 micromol/L at 42 hours or > 0,2 micromol/L at 66 hours after initiation of the methotrexate infusion. | From 36-66 hours after the initiation of methotrexate infusion.

SECONDARY OUTCOMES:
Development of methotrexate induced nephropathy, defined by an increase in serum creatinine by 50% or more compared with the serum creatinine concentration before start of each methotrexate infusion. | From the initiation of methotrexate infusion until 66 hours after.
Days of hospitalization in relation to the methotrexate infusion. | Days in relation to the methotrexate infusion and side effects.
Difference in baseline creatinine to highest serum creatinine between groups. | From initiation of the methotrexate infusion and up til 14 days after.
Drug exposure measured by area under the curve. | From 23 hours til 66 hours after initiation of the methotrexate infusion.
Duration and degree of side effects to the methotrexate treatment. | From initiation of the methotrexate infusion and up til on month after.
Total dosage of leucovorin. | From initiation of the methotrexate infusion and til serum methotrexate concentration is below 0,2 micromol/l.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Schrøder, MD, Study Director
Locations (1):
- Aarhus University Hospital, Skejby, Aarhus, Aarhus N, Denmark